CLINICAL TRIAL: NCT05785442
Title: Immunotherapy Navigated by Serum Presepsin for Infections of the Respiratory Tract: the INSPIRE Double-blind, Randomized, Phase IIa Exploratory Trial.
Brief Title: Use of Presepsin as a Marker for Immunotherapy Administration in Pneumonia
Acronym: INSPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INSPIRE; 2022-002390-28 (EudraCT Number)
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2023-09

CONDITIONS: Community-acquired Pneumonia; Hospital-acquired Pneumonia
Keywords: sepsis; presepsin; pneumonia; anakinra; SOFA
MeSH Terms: conditions — Community-Acquired Pneumonia; Healthcare-Associated Pneumonia; Sepsis; Pneumonia | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, double-blind, randomized, placebo-controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is designed to maintain blinding from participants, site investigators and their teams until completion of the study. At each center, there will be an unblinded pharmacist (and one substitute) who will be in charge of randomizing and preparing the study drug for each participant according to the randomized intervention assignment. These pharmacists will not be involved in data acquisition, collection, adjudication of outcomes or adverse events, or any other study procedures. They will not disclose the treatment assignment to the study team members unless it is via a formal process of early unblinding as described below.
  Αn independent biostatistician will generate the assignment to blinding treatment.
  Under normal circumstances, all the treatment assignments of participants will remain blinded until the completion of the trial (completion of enrollment and follow-up or early termination of the trial).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Treatment Arm 1: patients receiving placebo (N/S 0.9% w/v) subcutaneously once daily for 10 days plus Standard of Care
  Interventions: Drug: Placebo
- Anakinra (Active Comparator): Treatment Arm 2: patients receiving anakinra subcutaneously 100 mg once daily for 10 days plus Standard of Care
  Interventions: Drug: Anakinra Prefilled Syringe

INTERVENTIONS:
Drug: Anakinra Prefilled Syringe — Anakinra 100 mg administration subcutaneously once daily for 10 days (at least 4 days)
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebo — 0.67 ml N/S 0.9% w/v administration subcutaneously once daily for 10 days (at least 4 days)
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
The current study is an exploratory, phase IIa randomized clinical trial (RCT) aiming to evaluate if early presepsin increase coupled with early initiation of anakinra as an adjunct therapy to the standard-of-care treatment may improve outcomes of community-acquired pneumonia or hospital-acquired pneumonia.

DETAILED DESCRIPTION:
Sepsis is a potentially lethal syndrome, which is characterized by the dysregulated response of the host to an infection. Due to its severity, sepsis should always be considered in patients with confirmed or suspected infection as it can rapidly progress to organ failure with poor prognosis. Conversely, patients with new-onset organ failure should be suspected for occult infection. Current epidemiology is suggesting an increase in the incidence of new cases. Sepsis has considerable economic burden on the community as septic patients merit higher-level of healthcare and prolonged hospital stay. Subsequently, prompt recognition and treatment are of essence in order to mitigate the overall toll.

In the past years, numerous efforts have been made to identify a biomarker that portends the presence of sepsis, but none has managed to consistently predict which patients will eventually develop this syndrome. This is largely attributed to still-unknown host and pathogen mechanisms by which the sepsis cascade is initiated. Therefore, further understanding of the pathophysiology is of paramount importance.

The pathogenesis of sepsis is multifaceted and includes immune, cardiovascular, coagulation and metabolic perturbations. Immune dysregulation is a well-established component that leads to tissue injury. Activation of the innate immunity is a crucial step in the sequence of the upcoming events. As such, if we manage to early recognize the activation of one specific immune pathway during the initial stages of sepsis in the human host and promptly commence immunotherapy directed against this specific pathway, we may prevent the cascade of events leading the patient to life-threatening organ dysfunction. This paradigm of timely intervention on the immune system upon early recognition of a specific pathway activation is the SAVE-MORE trial in COVID-19. Preemptive initiation of anakinra treatment guided by the early increase of the biomarker suPAR (soluble urokinase plasminogen activator receptor) well before clinical signs of deterioration develop led to a 64% overall improvement and a 55% relative decrease in mortality. This early personalized treatment was registered in December 2021 by the European Medicines Agency.

One similar cascade of events is happening in sepsis. Bacterial lipopolysaccharide (LPS) of the cell membrane of Gram-negative bacteria and danger-associated molecular patterns (DAMPs) like high-mobility group box-1 (HMGB1) and mitochondrial DNA (mtDNA) are recognized by toll-like receptors (TLRs). Cluster of Differentiation 14 (CD14) is the naturally occurring receptor of LPS on the surface of monocytes/macrophages and the regulator of TLR-4 signal transduction. In 2004, a novel form of CD14, named soluble CD14 subtype (sCD14-ST) or presepsin was found significantly increased in patients with sepsis. Numerous studies have validated its use as an early indicator of sepsis, but a definite cut-off value has not been established due to the heterogeneity in the study design, selection of patients and clinical context. Once LPS binds and activates TLR-4, production of interleukin (IL)-1 ensues. As a consequence, early detection of increased presepsin coupled with anakinra, one short half-life inhibitor of the activity of IL-1α and IL-1β, may be a promising personalized treatment strategy for sepsis.

In recent years, studies conducted by the Hellenic Sepsis Study Group have shown that presepsin levels over 350 pg/ml have satisfactory diagnostic and prognostic value for sepsis. In particular, results from the INTELLIGENCE-1 study showed that in patients with at least one of the qSOFA criteria, presepsin more than 350 pg/ml has a sensitivity for diagnosing sepsis and 28-day mortality of 80.2% and 91.5%, respectively. Similar results were reproduced by 2 more independent studies; INTELLIGENCE-2, which also included patients with qSOFA ≥ 1 and SAVE trial, which investigated patients with COVID-19.

On the other hand, presepsin's role in determining the appropriateness of treatment remains unclear. In a controlled clinical trial conducted by Hongli Xiao et al, presepsin was used at predefined cut-offs in order to modulate the duration of antimicrobial therapy in septic patients. The primary endpoints were the number of days free of antibiotics in a 28-day period and mortality on days 28 and 90. The results revealed significantly fewer days of antibiotic exposure to the presepsin group (14.54 days vs. 11.01 days; P < 0.001).

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years
* Male or female gender
* In case of women of reproductive age, willingness to use dual contraceptive method during the study period
* Written informed consent provided by the patient. For subjects without decision-making capacity, informed consent must be obtained from a legally designated representative following the national legislation in the Member State where the trial is planned
* Community-acquired pneumonia or hospital-acquired pneumonia
* qSOFA score equal to 1
* Serum presepsin > 350 pg/ml

Exclusion Criteria:

* Age below 18 years
* Denial of written informed consent
* Any stage IV malignancy
* Any do not resuscitate decision
* Patients with PaO2/FiO2 less than 150 necessitating non-invasive ventilation or mechanical ventilation
* Hospitalization in Intensive Care Unit
* Known hypersensitivity to anakinra
* Oral or IV intake of corticosteroids at a daily dose equal to or greater than 0.4 mg/kg prednisone for a period greater than the last 15 days
* qSOFA score 0, 2 or 3
* Any anti-cytokine biological treatment for the last one month
* Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study
* Participation in any other interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Change of Sequential Organ Failure Assessment score by day 7 or death by day 90. | 90 days
  Patients who meet any of the following are considered to meet this endpoint: i) increase of Sequential Organ Failure Assessment score by 2 or more points from day 1 (before start of the study drug) until day 7; ii) death by day 90. Higher scores of the Sequential Organ Failure Assessment score indicate worsening of organ function, where the lowest score is 0 and highest is 24 (death).

SECONDARY OUTCOMES:
Change of Sequential Organ Failure Assessment score | 28 days
  Change of Sequential Organ Failure Assessment score over all days of follow-up. Higher scores indicate worsening of organ function, where lowest score is 0 and highest is 24 (death).
28-day organ dysfunction | 28 days
  Incidence of specific organ dysfunction by day 28
Time to hospital discharge | 28 days
  Time until discharge from hospital
28-day mortality | 28 days
  Mortality by day 28
90-day mortality | 90 days
  Mortality by day 90
Time to inflammation discontinuation | 7 days
  Time until attenuation of sepsis-induced inflammation as defined by procalcitonin measurements
Concentration of presepsin | 10 days
  Change of concentration of presepsin from baseline until day 10
Change in concentration of cytokines | 7 days
  Comparison of change of cytokine function by measurement of macrophage-derived, Th-1, Th-2 and Th-17 - derived cytokines' concentration following stimulation of cultured peripheral blood mononuclear cells (PBMCs). The concentrations of these molecules will be measured by enzyme-linked immunosorbent assay (ELISA) on days 1, 4 and 7.
Concentration of endothelial dysfunction markers | 7 days
  Comparison of change of endothelial dysfunction markers from baseline by days 4 and 7 by measurement of Intercellular Adhesion Molecule 1 (ICAM-1), Vascular Cell Adhesion Molecule 1 (VCAM-1), and E-selectin concentrations by enzyme-linked immunosorbent assay (ELISA).
Change of Sequential Organ Failure Assessment score of screening failure subjects | 10 days
  Comparative progression into overall organ dysfunction by day 10 (defined as in the primary endpoint) between patients who failed screening because of presepsin 350 pg/ml or less and patients who were enrolled in the study and were allocated to Treatment Arm 1 (placebo).
28-day mortality of screening failure cases compared with placebo | 28 days
  Comparative 28-day mortality between patients who failed screening because of presepsin 350 pg/ml or less and patients who were enrolled in the study and were allocated to Treatment Arm 1 (placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD, PhD, Study Chair — Hellenic Institute for the Study of Sepsis
Locations (5):
- Greece (5):
  - 4th Department of Internal Medicine, "Attikon" University Hospital, National and Kapodistrian University of Athens, Medical School, Athens
  - 1st Department of Internal Medicine, General Hospital of Athens GENNIMATAS, Athens
  - 1st Department of Internal Medicine, General Hospital of Eleusis THRIASIO, Athens
  - 6th Department of Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseases of Athens, Athens
  - 3rd Department of Internal Medicine, General Hospital of Nikaia AGIOS PANTELEIMON, Nikaia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tavoulareas G, Kontakou-Zoniou O, Antonakos N, Tasouli E, Adamis G, Kakavoulis N, Michelakis E, Skopelitis I, Dakou K, Psarrakis C, Koufargyris P, Astriti M, Sympardi S, Giamarellos-Bourboulis EJ. Efficacy of anakinra in reducing progression to organ dysfunction in patients with pneumonia (INSPIRE): a randomised, double-blind, placebo-controlled, phase IIa trial. Lancet Reg Health Eur. 2025 Dec 29;62:101573. doi: 10.1016/j.lanepe.2025.101573. eCollection 2026 Mar. PMID 41552367